CLINICAL TRIAL: NCT00141089
Title: Assessment of Efficacy and Safety of Tegaserod in Male Patients With Chronic Constipation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919E2309
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Constipation
Keywords: Male patients, chronic constipation, tegaserod
MeSH Terms: interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Tegaserod (HTF919) is an aminoguanidine indole compound and a member of a class of subgroup-selective 5-hydroxytryptamine (5-HT) agonists.

The aim of this study was to evaluate the efficacy and safety of tegaserod on bowel habits in male patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* A 6-month history of constipation defined as <3 complete spontaneous bowel movements per week and >1 of the following symptoms >25% of the time: hard stools, sensation of incomplete evacuation and straining

Exclusion Criteria:

* Patients with cancer, inflammatory bowel disease or other structural bowel disease
* Past or current diagnosis of irritable bowel syndrome were excluded.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1026
Dates: Start 2004-03; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with mean increase of more than one complete spontaneous bowel movement (csbm) per week during the first 4 weeks of treatment compared to baseline.

SECONDARY OUTCOMES:
For csbm and sbm : Increase of > or = of one/week for weeks 1 to 12 and week 1, absolute number for week 1 to 4 and 1 to 12, time to 1st csbm, sbm.
Daily assessment of bowel habits, patients assessment of bowel habits, constipation, distention/bloating, abdominal discomfort/pain, patients assessment of impact of constipation on quality of life, laxative use.
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Basel